CLINICAL TRIAL: NCT07277608
Title: Clinical Characteristics and Molecular Mechanism of Patients With Obstructive Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Zhaohui Tong, professor, Beijing Chao Yang Hospital
Other Study IDs: 2023-ke-450
Record Dates: First submitted 2024-01-03; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe OSA
- Non-severe OSA
- Healthy controls

SUMMARY:
To clarify the clinical features of patients with obstructive sleep apnea; To construct a multi-omics database of patients with obstructive sleep apnea, and compare the effects of different degrees of sleep apnea on prognosis, immunity, and metabolism. The medium and long-term prognosis, complications, comorbidities, risk factors, and immune and metabolic dynamics of patients with sleep apnea after treatment were studied. To elucidate the biomarkers and therapeutic targets associated with obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected obstructive sleep apnea (OSA) admitted to the sleep center of the respiratory Department of Beijing Chaoyang Hospital, Capital Medical University.
* Volunteer to participate in the study and sign an informed consent, and can complete at least 1 year of follow-up.

Exclusion Criteria:

* Patients with obstructive sleep apnea who have been treated with impermanent positive pressure ventilation;
* Pregnant or lactating women;
* Patients with severe respiratory failure requiring mechanical ventilation;
* Patients with severe heart, lung, liver, kidney, and central nervous system damage;
* Refuse to participate in follow-up visits and/or take biological samples.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with obstructive sleep apnea.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2033-08-07 (Estimated); Study Completion 2033-08-07 (Estimated)

PRIMARY OUTCOMES:
Multiple-omics features | Within 24 hours of admission，and samples of patients receiving treatment were also collected six months and one year after treatment
  ELISA ,proteomics and metabolomics were performed on blood, saliva, urine

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available on reasonable request.